CLINICAL TRIAL: NCT01865344
Title: A Pilot Study for the PainMonitor During Standardized Painful Stimuli and no Stimuli to Calculate the Sensitivity and Specificity and Thereby the Accuracy of the Monitor
Brief Title: Skin Conductance Fluctuations Per Sec and NRS to Monitor Pain
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Other Study IDs: REK sør-øst 2013/196
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Heart surgery: Pain monitoring at different time periods

SUMMARY:
To provide a preliminary evaluation of the correlation between Numeric rating Score (NRS) and skin conductance responses per second at rest and in response to a painful stimulus. Sensitivity and specificity will be calculated for NRS and skin conductance responses per sec to a standardized painful stimulus. Furthermore, predictors of pain will be examined.

DETAILED DESCRIPTION:
Cardiac surgery patients will be consented for participation in this trial. They will be asked about their pre-existing pain, anxiety about the needle-insertion and anxiety about the outcome of the operation, and employment status. This information will be obtained from self-reported schemas from the patients about presence/absence of pain and anxiety (the response options: yes/no) (1). The intensities of pain and anxiety will measured with NRS also ranging from 0 to 10 with one statement in each range: 0 no pain and 10 worst possible pain, and 0 no anxiety and 10 worst possible anxiety. The participants were requested to mark the point at the line that best agreed with how the pain and anxiety were experienced. The intensity of pain scored more than 3 on NRS was considered to be equal to moderate pain or more (1). Furthermore, patients in the Cardiac Surgery unit will be observed when undergoing pre-defined standardized painful stimuli as part of the standard of care treatment prior to and during surgery. The proposed study is structured using three events.

* Event 1: no stimuli, the period before placement of an arterial catheter when the patient has been administered diazepam, but is awake and calm. The registration will be for 1 min, 1 min before anticipated arterial line placement.
* Event 2: standardized painful stimulus, arterial catheter placement, with diazepam as premedication. The registration will be during arterial catheter placement.
* Event 3: no stimuli; patient is anesthetized before intubation. The registration will be for 1 min 1 min before anticipated intubation.
* There will also be one skin conductance response per sec registration for 1 min and the NRS score, one day postoperatively, when asking the patient about any side effects from the study.

During all defined events, the subject's skin conductance responses will be evaluated using the PainMonitor, and the subject will be asked to report pain using the 10 point NRS scale when awake. Before intubation when the patient is anesthetized, without stimuli, it is defined that the patient has no pain.

During these events, the number of skin conductance responses/sec will be analyzed in the defined time period, and this value will be used for statistical analyses. NRS scores will be obtained after the event and the value of the felt pain during the event will be asked for.

ELIGIBILITY:
Inclusion Criteria:

* Age: Older than 18 years, patients scheduled for cardiac surgery.
* Patients admitted to the Cardiac Unit with cardiac disease.
* Patients able to verbally communicate pain level during or after the procedures.
* Pain medication following institutional standard care; only diazepam given before the painful procedure. During surgery, institutional standard care for sedation will be given.

Exclusion Criteria:

* Administration or anesthesia or analgesia other than diazepam prior to evaluation with the PainMonitor.
* Presence of any neurological disease affecting the peripheral nerves.
* Abuse of alcohol or illicit drugs
* History of mental retardation or any mental disease
* Severe neuropathic disease
* Use of neostigmine before event 1, 2, and 3, see events below.
* Use of atropin
* Use of regional anesthesia at the extremity where the device electrodes are placed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cardiac patients prior to, during, and after anesthesia for surgery. The proposed pilot study will be conducted at the Acute Clinic, Rikshospitalet - Oslo University hospital, Oslo, Norway.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Skin conductance responses per sec and NRS before and during painful procedures | 8 months
  * No significant adverse events related to use of the Pain Monitor device
  * Increase in skin conductance responses per sec and NRS after administration of painful stimulus compared to the non-painful situations.

CONTACTS AND LOCATIONS:
Overall Officials: Jan F Bugge, MD.PhD, Principal Investigator — Head of the Anesthesia Thorax department
Locations (1):
- Acute Clinic, Rikshospitalet - Oslo University hospital, Oslo, Norway